CLINICAL TRIAL: NCT00883766
Title: PCOS and IVF: A Comparison Between Standard Long Protocol Versus an Antagonist Protocol Starting on Day 1
Brief Title: Polycystic Ovary Syndrome (PCOS) and In Vitro Fertilization (IVF): A Comparison Between Standard Long Protocol Versus an Antagonist Protocol Starting on Day 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Fulvia Mancini, Departamento de Obstetricia, Ginecologia y Reproducción
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX002
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2010-10

CONDITIONS: Polycystic Ovary Syndrome; In Vitro Fertilization
Keywords: Polycystic Ovary Syndrome; GnRH Antagonist; Long Agonist Protocol; OHSS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Long agonist protocol (Active Comparator)
  Interventions: Other: Controlled ovarian hyperstimulation for IVF with a long agonist protocol
- Antagonist protocol (Experimental)
  Interventions: Other: Controlled ovarian hyperstimulation for IVF with an antagonist protocol

INTERVENTIONS:
Other: Controlled ovarian hyperstimulation for IVF with a long agonist protocol — Day 1 of 1st menstruation: OC for 18-21 days (Microdiol ®) + Metformin (Dianben ®) 850 x 2/day if: BMI>30, HOMA >3.8, G/I ratio <4.5
  Day 18-24 of cycle: Leuprorelin (Procrin ®) 0.1 s.c. for 14-21 days
  Day 1 of 2nd menstruation (=Day 1 COH cycle): Hormonal profile (FSH, LH, E2, Pg, T, SHBG), Ultrasonography to exclude cyst >10 mm
  Day 2of COH cycle: rFSH (Gonal F ®) 150 IU/day for 4 days; Leuprorelin (Procrin ®) 0.1 s.c. (and following days)
  Day 7 of COH (and following): Measure FSH, LH, E2, Pg + Ultrasound
  Day before HCG: stop rFSH
  Day HCG: measure FSH, LH, E2, Pg, administer 250 mcg Choriogonadotropin-alfa ( Ovitrelle®)
  Day of pick-up: Follicular fluid from 1st follicle to be centrifuged and stored at -20°C
  Day 7 after pick-up: ultrasound, patient evaluation.
  Day 14 after pick-up: HCG in blood
  Day 28 after pick-up: Ultrasound to visualize heart beat if pregnancy test positive
  (OC= oral contraceptive; COH= Controlled Ovarian Hyperstimulation)
  Arms: Long agonist protocol
Other: Controlled ovarian hyperstimulation for IVF with an antagonist protocol — Day 1 of pre COH-cycle: OC for 18-21 days (Microdiol ®) + Metformin (Dianben ®) 850 x 2/day if: BMI>30, HOMA >3.8, G/I ratio <4.5
  Day 3 of free-pill interval: Hormonal profile (FSH, LH, E2, Pg, T, SHBG), Ultrasonography to exclude cyst >10 mm
  Day 5 of free-pill interval (=Day 1 COH cycle): Cetrorelix acetate (Cetrotide®) 0.25 mg s.c. + rFSH (Gonal F ®) 150 IU/day (and following days)
  Day 3-4-10 of COH cycle: measure FSH, LH, E2, Pg + ECO
  Day before HCG: stop rFSH + cetrorelix
  Day HCG: measure FSH, LH, E2, Pg, administer 250 mcg Choriogonadotropin-alfa ( Ovitrelle®)
  Day of pick-up: Follicular fluid from 1st follicle to be centrifuged and stored at -20°C
  Day 7 after pick-up: ultrasound, patient evaluation.
  Day 14 after pick-up: HCG in blood
  Day 28 after pick-up: Ultrasound to visualize heart beat if pregnancy test positive (OC= oral contraceptive; COH= Controlled Ovarian Hyperstimulation)
  Arms: Antagonist protocol

SUMMARY:
The aim of this study is to compare two different IVF-stimulation protocols in patients affected by PCOS: the use of a Gonadotropin-releasing hormone (GnRH) - antagonist starting on day 1 of controlled ovarian hyperstimulation (COH) versus a standard long agonist protocol; in order to assess whether it affects the number and quality of Metaphase II (MII) oocytes while reducing the risk of hyperstimulation. Since PCOS patients are also likely to be insulin resistant we also aim to evaluate how metformin affects tha IVF stimulation outcome.

DETAILED DESCRIPTION:
Hejinen et al (1) recently conducted a meta-analysis to compare outcomes of conventional IVF in women presenting with polycystic ovary syndrome (PCOS) and non-PCOS patients. They compared nine RCTs reporting data on 458 PCOS patients (793 cycles) and 694 matched controls (1116 cycles) and concluded that in PCOS there is an increased cancellation rate, but more oocytes retrieved per pick-up and a lower fertilization rate. Overall, PCOS and control patients achieved similar pregnancy and live birth rates per cycle. The incidence of ovarian hyperstimulation syndrome (OHSS) after oocyte retrieval was rarely reported.

Our results are in accordance with this meta-analysis. Therefore, if the pregnancy and abortion rates in PCOS and controls do not differ, the main problem when dealing with PCOS in IVF is OHSS. This condition can be approached by using an antagonist instead of an agonist, by changing the kind of ovulation trigger and by co-treating patients with metformin.

* One of the currently debatable issues regarding the use of GnRH antagonists refers to the timing of GnRH antagonist initiation. A fixed protocol starting antagonist arbitrarily on Day 6 of stimulation has been used in all introductory comparative trials employing a daily antagonist administration (2). Following these trials, a flexible antagonist initiation by a follicle of 14-15 mm has been evaluated. Currently, initiation of antagonist in the early follicular phase in PCOS patients has been performed by Lainas and coll. (3) who treated patients with PCOS either with a long GnRH agonist scheme or a fixed day-1 GnRH antagonist protocol and concluded that initiation of GnRH antagonist concomitantly with recombinant FSH on day 1 is associated with an earlier follicular growth and a different hormonal environment during the follicular phase when compared with the long agonist protocol. This may lead to a reduction in the incidence of OHSS.
* Over the past 15 years, it has become increasingly recognized that insulin resistance is central to the pathogenesis of the PCOS (4). Metformin, a biguanide insulin-lowering agent, has been extensively investigated in the management of PCOS. Two recent systematic reviews (5, 6) demonstrated that metformin improves reproductive function of some women with PCOS. Metformin also appeared to improve the outcomes of ovulation induction therapies when combined with clomiphene and gonadotrophin. Tang et al. recently studied PCOS overweight patients undergoing IVF to whom they administered 850 mg bid or placebo 28 days prior to the stimulation (7). They concluded that short-term co-treatment with metformin for patients with PCOS undergoing IVF/ICSI cycles does not improve the response to stimulation but significantly improves the pregnancy outcome and reduces the risk of OHSS.

The aim of this study is to verify if using an antagonist the number and quality of MII oocytes is equal compared to a standard long agonist protocol while reducing the risk of hyperstimulation.

Outcome measures:

Primary endpoints:

* Oocytes MII Secondary endpoints
* Fertilization rates
* Pregnancy rates
* Miscarriage rates
* Incidence of OHSS

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients according to the Rotterdam consensus criteria
* Presence of both ovaries
* Absence of endometriomas detected at ultrasound
* FSH < 10 IU/L on day 3 of the cycle
* E2 < 80 pg/mL, and Pg < 1.6 ng/mL at initiation of stimulation

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing's syndrome
* Androgen-producing tumours
* Hyperprolactinaemia and thyroid dysfunction
* Age > 38 years
* Serum FSH levels > 10 mIU/ml

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of Oocytes MII retrieved per patient | 1 Day

SECONDARY OUTCOMES:
Fertilization rates | 24 hours after pick-up
Clinical pregnancy rates | 4 weeks after pick-up
Incidence of OHSS | From ovulation triggering to two weeks after pick-up

CONTACTS AND LOCATIONS:
Overall Officials: Fulvia Mancini, M.D. PhD, Principal Investigator — Department of Obstetric, Gynecology and Reproductive Medicine
Locations (1):
- Institut Universitari Dexeus, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Heijnen EM, Eijkemans MJ, Hughes EG, Laven JS, Macklon NS, Fauser BC. A meta-analysis of outcomes of conventional IVF in women with polycystic ovary syndrome. Hum Reprod Update. 2006 Jan-Feb;12(1):13-21. doi: 10.1093/humupd/dmi036. Epub 2005 Aug 25. PMID 16123051
- [Background] Al-Inany H, Aboulghar M. GnRH antagonist in assisted reproduction: a Cochrane review. Hum Reprod. 2002 Apr;17(4):874-85. doi: 10.1093/humrep/17.4.874. PMID 11925376
- [Background] Lainas TG, Petsas GK, Zorzovilis IZ, Iliadis GS, Lainas GT, Cazlaris HE, Kolibianakis EM. Initiation of GnRH antagonist on Day 1 of stimulation as compared to the long agonist protocol in PCOS patients. A randomized controlled trial: effect on hormonal levels and follicular development. Hum Reprod. 2007 Jun;22(6):1540-6. doi: 10.1093/humrep/dem033. Epub 2007 Mar 8. PMID 17347165
- [Background] Tsilchorozidou T, Overton C, Conway GS. The pathophysiology of polycystic ovary syndrome. Clin Endocrinol (Oxf). 2004 Jan;60(1):1-17. doi: 10.1046/j.1365-2265.2003.01842.x. No abstract available. PMID 14678281
- [Background] Costello MF, Eden JA. A systematic review of the reproductive system effects of metformin in patients with polycystic ovary syndrome. Fertil Steril. 2003 Jan;79(1):1-13. doi: 10.1016/s0015-0282(02)04554-5. PMID 12524053
- [Background] Moll E, van der Veen F, van Wely M. The role of metformin in polycystic ovary syndrome: a systematic review. Hum Reprod Update. 2007 Nov-Dec;13(6):527-37. doi: 10.1093/humupd/dmm026. Epub 2007 Sep 1. PMID 17767003
- [Background] Tang T, Glanville J, Orsi N, Barth JH, Balen AH. The use of metformin for women with PCOS undergoing IVF treatment. Hum Reprod. 2006 Jun;21(6):1416-25. doi: 10.1093/humrep/del025. Epub 2006 Feb 24. PMID 16501038
- See also: Related Info — http://www.dexeus.com